CLINICAL TRIAL: NCT00447785
Title: Etude Des déterminants Endocrinologiques Des Apports énergétiques et Fluides Des Patients Alcooliques en Cours de Sevrage
Brief Title: Endocrine Regulation of Energy and Fluid Supplies in Alcoholic Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Other Study IDs: nutrialcohol
Record Dates: First submitted 2007-03-14; First posted 2007-03-15 (Estimated); Last update posted 2007-03-15 (Estimated); Status verified 2007-03

CONDITIONS: Alcoholism
Keywords: alcoholism; nutrition; craving; energy supplies; water supplies
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is about the endocrine regulation of energy and fluid supplies in alcoholic patients. A large proportion of energy and fluid is supplied by alcohol beverages in alcoholic patients. In this study, we evaluated the importance of these supplies with a detailed questionnaire, a nutrition software that evaluated the importance of each macro- and micronutrients and correlated these values with several hormones such as Leptin, Insulin, Cortisol, Ghrelin, and PYY involved in the regulation of energy balance or AVP involved in the regulation of plasma osmolality

DETAILED DESCRIPTION:
This study was conducted in a stepwise manner : study of the energy supplies first, of water supplies next.

Interviews and samples were performed or collected at two times of alcohol withdrawal to evaluate the possibility of parallel changes in craving for alcohol, supplies and endocrine function.

ELIGIBILITY:
Inclusion Criteria:

* Alcoholic patients still under the effect of alcohol at entry

Exclusion Criteria:

* Other type of addiction

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2004-09

CONTACTS AND LOCATIONS:
Overall Officials: Roussaux Jean Paul, MD, PhD, Study Chair — Cliniques Universitaires St Luc, Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires St Luc, Brussels, Belgium